CLINICAL TRIAL: NCT06670014
Title: A Randomized, Parallel-Group, Assessor-Blind, Multi-Center, Non-Inferiority Pivotal Study to Evaluate the Efficacy and Safety of the Digital Therapeutics 'repeech' for the Post-Stroke Dysarthria.
Brief Title: Evaluate the Efficacy and Safety of the Digital Therapeutics Repeech for the Post-Stroke Dysarthria.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HAII corp.ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDKC00
Record Dates: First submitted 2024-10-22; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Post-stroke Dysarthria

STUDY DESIGN:
Intervention Model Description: This is a two-arm interventional study comparing the efficacy of 'repeech' application to a workbook-based treatment for post-stroke dyasarthria.
  * Treatment group: Participants in the treatment group will use the 'repeech' application for 4 weeks, with recommended usage of 5 days per week, for 30 to 60 minutes per session.
  * Control Group: Participants in the control group will use a workbook provided by the sponsor, due the lack of a standarized care protocol for dysarthria. The control group will be instructed to use the workbook with the same frequency and duration as the treatment group (5 days per week, 30 to 60 minutes per session).
Who Masked: Outcomes Assessor
Masking Description: The study includes three blinded speech-language pathologists (SLPs) who will evaluate the speech intelligibility, the primary outcome measure. These SLPs will be blinded to the group assignments (treatment or control) of the participants. Each SLP will independentlry assess the speech intelligibility of participants at three times points: baseline, post-treatment, and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 'repeech' Intervention Group (Experimental): Participants in this group will use the 'repeech' for treatment.
  Interventions: Device: repeech
- Control Group (Other): Participants in the control group will use a workbook provided by the sponsor for the treatment of dysarthria.
  Interventions: Other: Workbook

INTERVENTIONS:
Device: repeech — Participants in this group will use the repeech application for a period of 4 weeks, with recommended usage of 5 days per week for 30 to 60 minutes per session. A designated speech-language pathologist (SLP) will set individualized treatment goals and customize the content of the therapy sessions based on each participant's baseline assessment. The repeech intervention will be tailored to meet the specific needs of each participant to improve speech intelligibility and communication abilities.
  Arms: 'repeech' Intervention Group
Other: Workbook — Participants in the control group will use a workbook provided by the sponsor for the treatment of dysarthria, due to the lack of a standardized care protocol for this condition. The recommended usage is the same as the treatment group: 5 days per week, for 30 to 60 minutes per session over a period of 4 weeks. After each self-treatment session, participants will record their activities on a checklist to monitor adherence and ensure compliance with the study protocol.
  Arms: Control Group

SUMMARY:
The goal of this interventional study is to evaluate the efficacy and safety of a digital therapeutic (DTx) application, 'repeech', for the treatment of post-stroke dysarthria. The study aims to assess improvement in speech intelligibility in individuals affected by post-stroke dysarthria using the DTx intervention.

DETAILED DESCRIPTION:
This study will evaluate a digital therapeutic (DTx), 'repeech', designed to complement tradtional speech therapy by addressing challenges such as accessibility, frequency of sessions, and personalized feedback. The 'repeech' offers an at-home, customzied intervention, providing patients with more flexible and accessible therapy options. It also encourage greater patient engagement in their treatment and promotes self-care.

The study is designed to assess the efficacy of the 'repeech' in improving speech function, especially speech intelligibility in individuals with post-stroke dysarthria. The clinical trial will be conducted across multiple sites to gather comprehensive data on the intervention's effectiveness and usability.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 19 years of age or older.
2. Participants must be neurologically stable post-stroke, as determined by a qualified physician.
3. Participants must have dysarthria due to stroke, with a National Institutes of Health Stroke Scale (NIHSS) score 1 (mild) or 2 (moderate) for dysarthria.
4. participants must have a Korean-Modified Mini-Mental State Examination (K-MMSE) score of 26 or higher within 1 month prior to enrollment in the study.
5. Participants must have sufficient visual, auditory, langauge, and motor abilities to understand and follow the assessment procedures, as determined by the Principal Investigator.
6. Participants must be able to use general-purpose digital equipment and comfortable with using the digital therapeutics(DTx) platform for this study.
7. Participants must provide informed consent after receiving a thorough explanation of the study, including potential risks and benefits. They must understand and agree to follow the study protocol.

Exclusion Criteria:

1. Participants with sigificant structural problems affecting the oral cavity and cervial region that would hinder accurate assessment.
2. Participants diagnosed with dementia, including Alzheimer's disease, Vascular dementia, Dementia due to Central Nervous System(CNS) infections (e.g., HIV, syphilis), Creutzfeldt-Jakob disease, Pick's disease, Huntington's disease, Parkinson's disease.
3. Participants currently receiving treatment for dementia within 3 months prior to study screening.
4. Participants who are unable to read or write in the language of the study.
5. Participants with severe mental health conditions including severe depression, schizophrenia, alcohol addicsion, drug dependence.
6. Participants with a severe langauge disorder, as determined by the physician(MD), that would significantly hinder their abiity to use digital therapeutics platform.
7. Participants deemed by the MD as unable to use general-purpose digital equipment.
8. Participants with additional medical or social concerns that, in the opinion of the Prindipal Investigator(PI), would make their participation in the clinical trial unsuitable or pose siginficant risks.
9. Participants who decline to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Speech Intelligibility | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  Speech intelligibility refers to how well a listener can understand the participant's speech. Participants will read sentences specifically developed to assess speech intelligibility. The speech samples will be evaluated by three blinded speech-language pathologists (SLPs), who will independently assess the intelligibility of each participants speech using a scale of 0 to 100, where 0 represents completely unintelligible and 100 represents perfect intelligibility. The average score from the three evaluations will be used for analysis.

SECONDARY OUTCOMES:
Maximum Phonation Time (MPT) | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  Maximum Phonation Time (MPT) refers to the longest duration a participant can sustain a vowel sound (e.g., ah,ee, or oo) on a single breath. The participants will follow instructions provided by repeech, which will guide them to take a deep breath and produce the sounds ah, ee, or oo for as long as possible. The app will record the duration of those sound, which will be measured in seconds.
Diadochokinesis Test, DDK | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  DDK measures the speed and accuracy of repetitive speech movements, assessing the overall language execution abillity in individuals with dysarthria.
  Measurement:
  * Alternate Motion Rate (AMR): Number of syllables (/pa/,/ta/,/ka/) per second, with assessment of regularity and accuracy of articulation. The unit will be times per second.
  * Sequential Motion Rate (SMR): Number of syllable sequences (/pataka/) per second, with assessment of regularity and accuracy of articulation. The unit will be times per second.
Percentage of consonants correct, PCC | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  DDK is to assess the accuracy of consonant articulation during a standarized word reading task.
  The participants read aloud a list of 30 words fromo a repeech application. The word list includes 43 consonants and 10 signle vowels.
  Accuracy of consonant articulation is calculated based on the number of correctly pronounced consonants within the 30-word reading task.
Patient Health Questionnaire--9, PHQ-9 | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  The PHQ-9 is a self-administered questionnair used to assess the severity of depressive sypmtoms in primary care settings. The PHQ-9 consists of 9 questions. Participants complete the PHQ-9 through the repeech application.
Quality of life in the dysarthric speaker, QoL-DyS | Baseline, 4 weeks (post-treatment), 8 weeks (Follow-up)
  The QoL-DyS is a self-reported questionnaire designed to assess the overall quality of life in individuals with dysarthria. It specifically explores the impact of dysarthria-related communication difficulties on various aspects of daily life.
  The Korean version of the QoL-DyS comprises 40 questions organized into 4 categories. Each category includes 10 questions, with responses typically measured on a Likert scale.
  Participants complete the Korean version of the QoL-DyS through the repeech application.
Compliance | 4 weeks (post-treatment)
  Treatment group compliance is measured through repeech application usage logs, capturing daily login times, task completion, and voice recordings. Data is collected over a 4-week clinical trial period.
  Control group compliance is measured through a self-reported checklist where participants record the dates of workbook use and task completion rates. Data is collected over a 4-week clinical trial period.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Yongin Severance Hospital, Yongin, Gyeonggi-do
  - Ewha Womans University Mokdong Medical Center, Seoul
  - Ewha Womans University Seoul Medical Center, Seoul
  - KyunHee University Hospital, Seoul
  - National Rehabilitation Center, Seoul